CLINICAL TRIAL: NCT04646122
Title: "Predicting Glaucoma Progression With Optical Coherence Tomography Structural and Angiographic Parameters".
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Ahmed Ali Youssif, Assiut, Assiut University
Other Study IDs: Glaucoma Progression with Opti
Record Dates: First submitted 2020-11-15; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Optical Coherence Tomography Glaucoma
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Optical Coherence Tomography — Optical Coherence Tomography parameters

SUMMARY:
to predict of glaucoma progression. By imaging of the retinal nerve fiber layer RNFL, optic nerve head (ONH) and macular measurements using spectral-domain OCT (SD-OCT) instruments

,and detection of optic disc perfusion changes using OCTA.

DETAILED DESCRIPTION:
Subjects will go a comprehensive ophthalmologic examination including review of medical history, best-corrected visual acuity (BCVA), slit-lamp biomicroscopy, intraocular pressure (IOP) measurement, gonioscopy, dilated fundoscopic examination, stereoscopic optic disc photography, and automated perimetry using Swedish Interactive Threshold Algorithm (SITA Standard 24-2). Only subjects with open angles on gonioscopy were included.

One eye of each subject will be scanned by a high-speed 1050-nm-wavelength swept-source OCT instrument.

OCT is providing measurements of the RNFL thickness, ONH, as well as the inner macula for the assessment of glaucoma progression.

The split-spectrum amplitude-decorrelation angiography (SSADA) algorithm will be used to compute 3-dimensional optic disc angiography. A disc flow index was computed from 4 registered scans.

Evaluation of progressive changes of the optic disc and RNFL will be based on event-analysis and/or trend-analysis. In event analysis, progression is defined when the difference between the baseline and follow-up measurements of the parameter of interest is greater than its test-retest variability (or the reproducibility coefficient). In trend analysis, regression analysis is performed between the parameter of interest and time.

ELIGIBILITY:
1. Inclusion criteria:

   * Patients older than 18 years of age with primary open-angle glaucoma (OAG) .
   * Primary OAG (POAG) diagnosed on the basis of IOP measurements more than 21 mmHg, open angle on gonioscopy (Grade 3 or 4 on Schaffer grading system for angle width), glaucomatous visual field defects consistent with glaucomatous optic disc changes.
   * Eyes with baseline macular and ONH OCT images and ONH photographs of adequate quality and r performed within 6 months of each other were selected
2. Exclusion criteria:

   * Participants with significant retinal disease.
   * non-glaucomatous optic neuropathy.
   * anomalous discs
   * any retinal pathology. A history of cataract or glaucoma surgery will not be exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will go a comprehensive ophthalmologic examination including review of medical history, best-corrected visual acuity (BCVA), slit-lamp biomicroscopy, intraocular pressure (IOP) measurement, gonioscopy, dilated fundoscopic examination, stereoscopic optic disc photography
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
retinal nerve fiber layer RNFL | one year
  Thickness using OCT
optic nerve head (ONH) | one year
  Thickness using OCT

SECONDARY OUTCOMES:
disc perfusion changes | one year
  flow index using OCTA

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Fathallah, Phd, Study Director — Assiut University

REFERENCES:
- [Background] Bussel II, Wollstein G, Schuman JS. OCT for glaucoma diagnosis, screening and detection of glaucoma progression. Br J Ophthalmol. 2014 Jul;98 Suppl 2(Suppl 2):ii15-9. doi: 10.1136/bjophthalmol-2013-304326. Epub 2013 Dec 19. PMID 24357497
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940